CLINICAL TRIAL: NCT01325077
Title: Efficacy of a Nurse-based, Anesthesiologist-supervised Acute Pain Service for Pediatric Patients
Acronym: Nurse-APS
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Professor Suwannee Suraseranivongse, Faculty of Medicine Siriraj hospital, Mahidol University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Si 603/2010; 545/2553(EC3) (Registry Identifier: 545/2553(EC3))
Record Dates: First submitted 2011-03-06; First posted 2011-03-29 (Estimated); Last update posted 2011-03-29 (Estimated); Status verified 2011-03

CONDITIONS: Postoperative Pain; Satisfaction
Keywords: Nurse-based, acute pain service, pediatric, postoperative,; pain
MeSH Terms: conditions — Pain, Postoperative; Personal Satisfaction; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Conventional model, Study model (Experimental): Conventional model(C): Nurses give fixed-dose analgesic according to surgeons' prescription Study model(S): Nurses give initial-dose analgesic according to surgeons' prescription. In case of inadequate pain relief, another half of initial dose will be given twice at 15-min interval and acute pain service will be consulted if there is still pain.
  Interventions: Other: model of health care service

INTERVENTIONS:
Other: model of health care service — Conventional model(C): Nurses give fixed-dose analgesic according to surgeons' prescription Study model(S): Nurses give initial-dose analgesic according to surgeons' prescription. In case of inadequate pain relief, another half of initial dose will be given twice at 15-min interval and acute pain service will be consulted if there is still pain.

SUMMARY:
Can a nurse-based, anesthesiologist-supervised model reduce prevalence of postoperative pain in pediatric patients?

DETAILED DESCRIPTION:
Comparison of 2 treatment model in reducing prevalence of postoperative pain in pediatric patients:

Conventional model(C): Nurses give fixed-dose analgesic according to surgeons' prescription Study model(S): Nurses give initial-dose analgesic according to surgeons' prescription. In case of inadequate pain relief, another half of initial dose will be given twice at 15-min interval and acute pain service will be consulted if there is still pain.

ELIGIBILITY:
Inclusion Criteria:

* Age up to15 years old
* Underwent surgery with moderate to severe pain

Exclusion Criteria:

* ENT, Eye, ambulatory surgery
* Cardiac, Neurosurgery
* Severe neurocognitive impairment
* Continuous epidural analgesia which anesthesiologists take care by themselves

Ages: 31 Days to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 103 (Estimated)
Dates: Start 2011-03; Primary Completion 2011-10 (Estimated); Study Completion 2011-10 (Estimated)

PRIMARY OUTCOMES:
prevalence of patients with moderate to severe pain more than once in first postoperative day | 24 hours
  moderate to severe pain = Neonatal Infant Pain Scale =,>4 or CHEOPS =,>8 or Verbal numerating scale =,>4

CONTACTS AND LOCATIONS:
Overall Officials: Suwannee Suraseranivongse, MD, Principal Investigator — Mahidol University
Locations (1):
- Departnment of Anesthesiology,Siriraj Hospital, Mahidol University, Bangkok, Thailand